CLINICAL TRIAL: NCT06099860
Title: Therapeutic Impact of Kinesio Taping Along With Balance Training in Patients With Chronic Low Back Pain of Sacroiliac Joint Dysfunction:A Randomized Control Study
Brief Title: Therapeutic Impact of KT Along With BT in Patients With Chronic Low Back Pain of Sacroiliac Joint Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Najran University (Other)
Responsible Party: Principal Investigator, Hashim Ahmed, Assistant Professor, Najran University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IE/IIMS&R/2022/78
Record Dates: First submitted 2023-10-19; First posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Sacroiliac Joint Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): KBT Group
  Interventions: Other: Kinesio Taping; Other: Balance Training (BT); Other: Hot Pack and Stretching Exercises
- Group B (Experimental): BT Group
  Interventions: Other: Balance Training (BT); Other: Hot Pack and Stretching Exercises

INTERVENTIONS:
Other: Kinesio Taping — Kinesio tape with a 5 cm width was used. Participants were positioned on the side lying on the non-involved side with the hip joint of the involved side flexed to 45 degrees and the femur supported in neutral rotation. First, the tape was placed over the area between the ASIS and PSIS to protect the skin. Next, two strips of tape were applied over the first tape to correct anterior innominate rotation. The first piece was applied at the ASIS and pulled firmly to the PSIS in a straight anterior-to-posterior direction. The second piece was applied in an arching manner pulled firmly from the ASIS to the PSIS. the tape was changed once every 3 days
  Arms: Group A
Other: Balance Training (BT) — The balance training was performed on the Biodex balance system, participants wwere instructed to stand on a podium and stabilize themselves to keep the cursor in the middle of co-centered circle on the displayed screen/monitor. Stability level of platform was set on eight for first two sessions and then reduced to one level on every two sessions so that in the 9th and 10th session the stability level was four. From session four onwards, the participants performed the limit of stability exercises with Biodex Balance System. The participants performed this exercise protocol two times in each session. Total 12 sessions were given in time period of six weeks.
Other: Hot Pack and Stretching Exercises — A hot pack was applied for 20 minutes, stretching exercises were performed.

SUMMARY:
This research aimed to determine the impacts of KT and balance exercises in patients with CLBP of SIJ dysfunction.

DETAILED DESCRIPTION:
The study will be based on a two-arm parallel group randomized control design. thirty participants of CLBP of SIJ Dysfunction will be recruited from the Physiotherapy department, at Integral University, India. Study objectives and procedure will be properly explained and written informed consent will be obtained at the beginning of the study. All the participants will be randomly divided into two groups A and B. Experimental group A will receive the hot pack, Stretching exercise, and Kinesio taping along with balance training (KBT), and group B will receive the hot pack, Stretching exercise, and Balance training (BT) exercise

ELIGIBILITY:
Inclusion Criteria:

* Subjects having chronic (>3 months) non-specific low back pain (NSLBP) of sacroiliac joint (SIJ) origin
* Age 20-50 years.
* Presence of pain exacerbated as a result of bending laterally or backward.
* Positive results on at least 2 of the pain-provocation tests [FABER, Posterior shear, and Gaenslen pain provocation tests) and one of the motion palpation tests (ie, Gillet and forward flexion tests) .

Exclusion Criteria:

* past or current history of surgery or major trauma to spine, pelvis, lower limb, chest or abdomen in the past 12 months.
* lower extremity musculoskeletal disorders.

  .localized spinal pathology, congenital anomalies of hip, pelvis or spine that limits mobility -systematic arthropathy, neuropathy or metabolic disorder
* Presence of other causes of LBP such as lumbar discopathy and spinal stenosis discovered via clinical examination and MRI scanning
* pregnancy.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-10-12 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | 6 Weeks
  Pain intensity was measured by using the Visual Analog Scale (VAS), a linear scale wherein patients indicate their pain intensity on a 10 cm line ranging from 'no pain' to 'worst imaginable pain'
Functional disability | 6 Weeks
  Functional disability was measured by using the Oswestry Disability Index (ODI), a validated 10-item questionnaire evaluating various dimensions of daily living
Balance | 6 Weeks
  The balance was measured by using the Biodex Balance System (BBS).overall (OA), the anteroposterior (AP), and the mediolateral (ML) stability scores were measured.

CONTACTS AND LOCATIONS:
Overall Officials: Hashim Ahmed, PhD, Principal Investigator — Najran University
Locations (1):
- Integral University Hospital, Lucknow, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: No